CLINICAL TRIAL: NCT04802343
Title: A Single-center, Randomized, Placebo-controlled, Parallel-group, Double-blind Study to Investigate the Pharmacokinetics, Safety and Tolerability of Single and Multiple Oral Doses of BAY 1817080 in Chinese Healthy Adult Male Participants.
Brief Title: A Trial to Learn How BAY1817080 Moves Into, Through and Out of the Body and How Safe it is in Healthy Chinese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: 21009
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics (PK)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY1817080 dose escalation (Experimental): Healthy male subjects will receive BAY1817080 dose 1 and dose 2 as a single oral dose and BAY1817080 dose 3 as a single oral dose on Day 1 and twice daily (BID) from Day 7 to Day 16 followed by a last dose in the morning of Day 17.
  Interventions: Drug: BAY1817080
- Placebo (Placebo Comparator): Healthy male subjects will received corresponding placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1817080 — Oral, tablet.
  Arms: BAY1817080 dose escalation
Drug: Placebo — Oral, tablet.
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat chronic cough. Before patients with medical conditions can join clinical trials, researchers do trials in healthy participants first to understand how the body acts on the new treatment and learn how safe it is.

In this trial, the researchers will study how much of the trial drug, BAY1817080, gets into the blood in a small number of participants. The trial will include about 39 healthy Chinese male who are aged 18 to 45.

For this trial participants will be divided in 3 groups. Groups 1 and 2 will take either dose 1 or dose 2 of BAY1817080 or placebo 1 time. Participants of groups 3 will take dose 3 of BAY1817080 or placebo one time at the first day and continue to take dose 3 of BAY1817080 twice a day from day 7 to day 16 of the trial. On day 17 they will take only one dose 3 of BAY1817080.

All participants will take BAY1817080 or a placebo as a tablet by mouth. For this trial, the participants in Groups 1 and 2 will stay at the trial site for up to 10 days. The participants in Group 3 will stay at the trial site for up to 26 days. The trial will last up to 4 weeks for the participants in Groups 1 and 2, and 6 weeks for the participants in Group 3.

During the trial, the doctors will take blood and urine samples and check the participants blood pressure, pulse rate and electrocardiogram (ECG). The participants will answer questions about how they are feeling to check their general wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy according to complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-Lead electrocardiogram (ECG), and clinical laboratory tests
* Race: Chinese
* Age: 18 to 45 years (inclusive) of age
* Weight: Body mass index (BMI): ≥ 18.0 and <= 27.9 kg/m²
* Male participants
* Subjects who agree to use adequate contraception when sexually active during the study period and for 90 days after receiving the investigational medicinal product and not to act as sperm donor for 90 days after dosing.

Exclusion Criteria:

Medical and Surgical History

* Any findings from the medical examination (including medical history, physical examination, vital signs, laboratory tests and ECG) deviating from normal and deemed by the investigator to be of clinical relevance
* Medical history of hypogeusia/dysgeusia or dysfunction in the ability to taste
* Any known presence or history of severe allergies, non-allergic drug reactions, or multiple drug allergies
* Known or suspected malignant tumors or carcinoma in situ
* Known liver disease: existing acute or chronic progressive liver disease, e.g. disturbance of bilirubin excretion (Dubin-Johnson and Rotor syndromes); disturbances of bile secretion and flow (cholestasis); presence or history of liver tumors (benign or malignant). (Note: According to this criterion, there must have been an interval of at least 6 months between the subsidence of any viral hepatitis [normalization of liver parameters] and the screening visit.)
* Any known relevant kidney disease (e.g. glomerulonephritis) or any renal injury associated with multisystem diseases/disorders (e.g. systemic lupus erythematosus, diabetic nephropathy)
* Known metabolic disorders (e.g. diabetes mellitus, severe hypertriglyceridemia)
* Known cardiovascular disorders requiring treatment
* Migraine with neurological symptoms (complicated migraine)
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known hypersensitivity to the study interventions including components of the preparation Medication, drug use and special behavioral patterns
* Regular use of therapeutic or recreational drugs, e.g. carnitine products, anabolics, high-dose vitamins
* Intake of drugs with a long half-life (>24 hours) within a timeframe of less than 5 half-lives before study drug administration
* Use of any systemic or topically active drug(s) that might influence the results of the study within the 14 days before study intervention administration or during the study until follow-up. (Note: This includes drugs that might affect the PK of BAY 1817080, e.g. laxatives, loperamide, metoclopramide, antacids, H2-receptor antagonists, cytochrome P450 [CYP] 3A4 inducers, strong CYP3A4 inhibitors).

Electrocardiogram, blood pressure, pulse rate

* Clinically relevant ECG findings, such as a second- or third-degree atrioventricular block, prolongation of the QRS complex over 120 msec at screening or pre-dose baseline measurement on Day -1 Physical examination
* Clinically relevant findings in the physical examination Neurological examination
* Clinically relevant findings in the orientating, basic neurological examination Laboratory examination
* Positive result in urine drug screening, or positive alcohol breath test Other
* Participation in another study and received an investigational drug within the 2 months or a longer and more appropriate time as determined by the investigator (e.g. approx. 5 half-lives of the previous investigational drug) before first study intervention administration
* Criteria that in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the participant's safety

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Cmax of BAY1817080 dose 1 and dose 2 (Day 1) | Pre-dose on Day 1 to 216 hours post-dose
  Cmax: maximum observed drug concentration in measured matrix after single dose administration
Cmax of BAY1817080 dose 3 (Day 1) | Pre-dose on Day 1 to 144 hours post-dose
  Cmax: maximum observed drug concentration in measured matrix after single dose administration
AUC of BAY1817080 dose 1 and dose 2 (Day 1) | Pre-dose on Day 1 to 216 hours post-dose
  AUC: area under the concentration vs. time curve
AUC of BAY1817080 dose 3 (Day 1) | Pre-dose on Day 1 to 144 hours post-dose
  AUC: area under the concentration vs. time curve
Cmax,md of BAY1817080 in dose 3 cohort (Day 17) | Pre-dose on Day 17 to 12 hours post-dose
  Cmax,md: maximum observed drug concentration in measured matrix after multiple dose administration during a dosage interval, directly taken from analytical data
AUCτ,md of BAY1817080 in dose 3 cohort (Day 17) | Pre-dose on Day 17 to 12 hours post-dose
  AUCτ,md: the area under the concentration-time curve in the dosing interval after multiple doses

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) with intensity | From the first dose of study intervention up to the follow-up visit (up to 30 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Li X, Haranaka M, Li H, Liu P, Chen H, Klein S, Reif S, Francke K, Friedrich C, Okumura K. P2X3 Receptor Antagonist Eliapixant in Phase I Clinical Trials: Safety and Inter-ethnic Comparison of Pharmacokinetics in Healthy Chinese and Japanese Participants. Clin Pharmacokinet. 2024 Jun;63(6):901-915. doi: 10.1007/s40262-024-01387-y. Epub 2024 Jun 21. PMID 38907175